CLINICAL TRIAL: NCT01296568
Title: Disposition of [14C]LY2603618 Following Intravenous Administration in Patients With Advanced and/or Metastatic Solid Tumors
Brief Title: C14 Study in Oncology Patients With Advanced and/or Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13525; I2I-MC-JMMH (Other: Eli Lilly and Company)
Record Dates: First submitted 2011-02-14; First posted 2011-02-15 (Estimated); Results first posted 2018-10-25 (Actual); Last update posted 2019-01-07 (Actual); Status verified 2018-12

CONDITIONS: Advanced Cancer
Keywords: metastatic solid tumors; Malignant/M-Neoplasm; Pancreas NOS; Absorption; Distribution; Metabolism; Excretion; Mass balance; Metabolic profile; Radiolabeled study
MeSH Terms: interventions — LY2603618; Pemetrexed; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LY2603618 (Experimental): Single 250 milligram (mg) intravenous dose of LY2603618 containing carbon-14-labeled LY2603618 ([^14C]LY2603618).
  After the completion of a minimum 7-day washout period, participants may receive additional doses of LY2603618 in combination as follows:
  * Gemcitabine 1000 milligrams per square meter (mg/m^2) on Days 1, 8, and 15 with 230 mg LY2603618 being administered on Days 2, 9 and 16 of a 28-day cycle OR
  * Pemetrexed 500 mg/m^2 on Day 1 and 275 mg LY2603618 on Day 2 of a 21-day cycle
  Participants will be allowed to continue to receive the combination therapy until fulfilling one of the criteria for discontinuation, such as unacceptable toxicity or disease progression.
  Interventions: Drug: LY2603618; Drug: Pemetrexed; Drug: Gemcitabine

INTERVENTIONS:
Drug: LY2603618 — Administered intravenously
Drug: Pemetrexed — Administered intravenously
  Other Names: LY231514; Alimta
Drug: Gemcitabine — Administered intravenously
  Other Names: LY188011; Gemzar

SUMMARY:
This is an open-label study being conducted to determine the metabolism and physiological disposition of radiolabeled LY2603618 after a single dose in patients with advanced and/or metastatic solid tumors.

After a minimum 7-day washout period following the carbon-14-labeled LY2603618 ([^14C]LY2603618) dose, patients will be allowed to continue to receive continued access to LY2603618 in combination with pemetrexed or gemcitabine as outpatients.

ELIGIBILITY:
Inclusion Criteria:

* Have a histological or cytological diagnosis of cancer (solid tumor), with clinical or radiologic evidence of locally advanced and/or metastatic disease, for which no life-prolonging therapy exists (that is, refractory to standard therapy and/or therapies known to provide clinical benefit, or for which no standard therapy exists). Note: participants who have had progressive disease after receiving pemetrexed for metastatic disease are excluded from receiving the combination with pemetrexed during the safety extension study. Participants who have had progressive disease after receiving gemcitabine for metastatic disease are excluded from receiving the combination with gemcitabine during the safety extension study.
* Have a body surface area greater than or equal to 1.37 meters squared (m^2)
* Have given written informed consent prior to any study-specific procedures
* Adequate hematologic, hepatic and renal function
* Have a performance status of less than or equal to 2 on the Eastern Cooperative Oncology Group (ECOG) scale
* Have discontinued all previous treatments for cancer, including chemotherapy, radiotherapy, anticancer hormone therapy, or other investigational therapy for at least 30 days prior to study entry and recovered from the acute effects of therapy (at least 42 days for mitomycin-C or nitrosoureas, or 60 days for monoclonal antibodies)
* Are reliable and willing to make themselves available for the duration of the study and are willing to follow study procedure
* Males and females with reproductive potential: Must agree to use medically approved contraceptive precautions during the study and following the last dose of study drug until, in the judgment of the investigator, it is safe for the participant to become pregnant or father a child
* Females with childbearing potential: Have had a negative serum pregnancy test less than or equal to 7 days before the first dose of study drug and must also not be breastfeeding
* Have an estimated life expectancy that, in the judgment of the investigator, will permit the participant to complete 1 full cycle of treatment (beyond the initial [^14C]LY2603618 dose)
* Prior radiation therapy for treatment of cancer other than pancreatic is allowed to <25% of the bone marrow and participants must have recovered from the acute toxic effects of their treatment prior to study enrollment. Prior radiation to the whole pelvis is not allowed. Prior radiotherapy must be completed at least 4 weeks before study entry.

Exclusion Criteria:

* Have received treatment within 28 days of the initial dose of study drug with an experimental agent for noncancer indications that has not received regulatory approval for any indication
* Have previously completed or withdrawn from this study or any other study investigating LY2603618 or any other checkpoint kinase one (Chk1) inhibitor
* Have a known allergy to gemcitabine, pemetrexed, LY2603618, or any ingredient of gemcitabine, pemetrexed, or LY2603618 (like Captisol)
* Have serious preexisting medical conditions (left to the discretion of the investigator) other than advanced cancer
* Have symptomatic central nervous system (CNS) malignancy or metastasis (screening not required). Participants with treated CNS metastases are eligible for this study if they are not currently receiving corticosteroids and/or anticonvulsants, and their disease is asymptomatic and radiographically stable for at least 90 days
* Have current hematologic malignancies or either acute or chronic leukemia
* Have an active fungal, bacterial, and/or known viral infection including human immunodeficiency virus (HIV) or viral (A, B, or C) hepatitis (screening is not required)
* Have a QTc interval of >500 milliseconds (msec) on the screening electrocardiogram (ECG)
* Have ECG abnormalities on the screening ECG such as significant conduction abnormalities, ischemic changes (such as prior Q-wave myocardial infarction and/or marked ischemic ST- and T-wave), arrhythmias (such as persistent or paroxysmal ventricular or supraventricular arrhythmias, including atrial fibrillation), or other ECG abnormalities that would put the participant at unnecessary risk in the opinion of the investigator
* Have participated in a ^14C study within the last 6 months prior to screening for this study. The total exposure from this study and the previous study must be less than 5 milliSieverts (mSv).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2011-02; Primary Completion 2011-12 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9AM-5PM Eastern time (UTC/GMT- 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bruderholz, Switzerland

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study had 2 phases. First phase: participants (pts) received single dose of carbon-14-labeled LY2603618 ([^14C]LY2603618) and completed a minimum 7-day washout. Second phase: pts had option to continue receiving LY2603618 in combination with gemcitabine or pemetrexed. All pts chose to receive gemcitabine for combination treatment.
Groups:
- Entire Study Population: In the [^14C]LY2603618 Single Dose and Washout Phase (first phase), participants received a single 250 milligram (mg) dose of LY2603618 containing [^14C]LY2603618, administered as a 1-hour intravenous infusion. Participants then completed a minimum 7-day washout period.
  In the Continued Access Phase (second phase), participants received additional doses of LY2603618 in combination with gemcitabine as follows:
  • Gemcitabine 1000 milligrams per square meter (mg/m^2) administered as an intravenous infusion on Days 1, 8, and 15 with 230 mg LY2603618 administered intravenously on Days 2, 9 and 16 of a 28-day cycle.
  Participants were allowed to continue to receive the combination therapy until fulfilling 1 of the criteria for discontinuation, such as unacceptable toxicity or disease progression.
Period: [^14C]LY2603618 Single Dose and Washout
Arm/Group | Entire Study Population
Started | 3
Completed | 3
Not Completed | 0
Period: Continued Access Phase
Arm/Group | Entire Study Population
Started | 3
Completed | 0 (After study discontinuation participants assessed for disease progression (21-day safety follow-up).)
Not Completed | 3
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 1
Not completed — Disease Progression | 1

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 3
Region of Enrollment [Count of Participants; unit: Participants]
  Switzerland | 3

OUTCOME MEASURES:

1. Primary Outcome: Urinary and Fecal Excretion of LY2603618 Radioactivity Over Time Expressed as a Percentage of the Total Radioactive Dose Administered
Description: Urinary and fecal excretion samples from each participant were measured by liquid scintillation counting. The radioactive counts detected in urine and fecal samples were each divided by the theoretical radioactive count in the total radioactive dose administered and multiplied by 100% to arrive at a percentage of total radioactive dose excreted in urine and feces.
Time Frame: 0 to 6 hours, 6 to 12, 12 to 24, 24 to 48, 48 to 72 and 72 to 96 hours post-dose
Population: All enrolled participants.
Measure: Mean (Standard Deviation); unit: percentage of total dose
Groups:
- [^14C]LY2603618: Participants in the first phase of the study received a single 250 milligram (mg) dose of LY2603618 containing [^14C]LY2603618, administered as a 1-hour intravenous infusion. Participants then completed a minimum 7-day washout period.
Arm/Group | [^14C]LY2603618
Number analyzed (Participants) | 3
percentage of total dose
  Feces | 72.2 (2.52)
  Urine | 11.0 (0.57)

2. Secondary Outcome: Plasma Pharmacokinetics of LY2603618: Maximum Observed Drug Concentration (Cmax)
Description: Plasma LY2603618 Cmax following a single dose on Day 1.
Time Frame: 0, 0.5, 1, 2, 4, 6, 8, 12, 24, 48, 72 and 96 hours post-dose
Population: All enrolled participants.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | [^14C]LY2603618
Number analyzed (Participants) | 3
nanograms per milliliter (ng/mL) | 4750 (52)

3. Secondary Outcome: Plasma Pharmacokinetics of Radioactivity: Maximum Observed Drug Concentration (Cmax)
Description: Plasma radioactivity Cmax [nanogram equivalents per milliliter (ng Eq/mL)] following a single dose on Day 1.
Time Frame: 0, 0.5, 1, 2, 4, 6, 8, 12, 24, 48, 72 and 96 hours post-dose
Population: All enrolled participants.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng Eq/mL
Arm/Group | [^14C]LY2603618
Number analyzed (Participants) | 3
ng Eq/mL | 5660 (47)

4. Secondary Outcome: Plasma Pharmacokinetics of LY2603618: Area Under the Concentration Time Curve From Time Zero to Infinity [AUC(0-infinity)]
Description: Plasma LY2603618 AUC(0-infinity) following a single dose on Day 1.
Time Frame: 0, 0.5, 1, 2, 4, 6, 8, 12, 24, 48, 72 and 96 hours post-dose
Population: All enrolled participants.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hours per milliliter (ng*h/mL)
Arm/Group | [^14C]LY2603618
Number analyzed (Participants) | 3
nanograms*hours per milliliter (ng*h/mL) | 22300 (48)

5. Secondary Outcome: Plasma Pharmacokinetics of Radioactivity: Area Under the Concentration Time Curve From Time Zero to Infinity [AUC(0-infinity)]
Description: Plasma radioactivity AUC(0-infinity) [nanogram equivalents*hours per milliliter (ng Eq*h/mL)] following a single dose on Day 1.
Time Frame: 0, 0.5, 1, 2, 4, 6, 8, 12, 24, 48, 72 and 96 hours post-dose
Population: All enrolled participants.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng Eq*h/mL
Arm/Group | [^14C]LY2603618
Number analyzed (Participants) | 3
ng Eq*h/mL | 32500 (63)

6. Secondary Outcome: Plasma Pharmacokinetics of LY2603618: Area Under the Concentration Time Curve From Time Zero to Time t [AUC(0-tlast)]
Description: Plasma LY2603618 AUC(0-tlast) where tlast is the last time point with a measurable concentration following a single dose on Day 1.
Time Frame: 0, 0.5, 1, 2, 4, 6, 8, 12, 24, 48, 72 and 96 hours post-dose
Population: All enrolled participants.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hours per milliliter (ng*h/mL)
Arm/Group | [^14C]LY2603618
Number analyzed (Participants) | 3
nanograms*hours per milliliter (ng*h/mL) | 22200 (48)

7. Secondary Outcome: Plasma Pharmacokinetics of Radioactivity: Area Under the Concentration Time Curve From Time Zero to Time t [AUC(0-tlast)]
Description: Plasma radioactivity AUC(0-tlast) [nanogram equivalents*hours per milliliter (ng Eq*h/mL)] where tlast is the last time point with a measurable concentration following a single dose on Day 1.
Time Frame: 0, 0.5, 1, 2, 4, 6, 8, 12, 24, 48, 72 and 96 hours post-dose
Population: All enrolled participants.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng Eq*h/mL
Arm/Group | [^14C]LY2603618
Number analyzed (Participants) | 3
ng Eq*h/mL | 27700 (56)

8. Secondary Outcome: Relative Abundance of LY2603618 and the Metabolites of LY2603618 in Urine
Description: Relative abundance was expressed as the percentage of the dose of study drug administered and calculated as %=[amount of LY2603618 or its metabolites excreted/amount of radioactive dose administered]*100.
Time Frame: Day 1 through 7 days postdose
Population: All enrolled participants.
Measure: Mean (Full Range); unit: percentage of [^14C]LY2603618
Arm/Group | [^14C]LY2603618
Number analyzed (Participants) | 3
percentage of [^14C]LY2603618
  LY2603618 (parent) | 3.3 [2.3 to 5.1]
  Metabolites | 3.0 [2.5 to 3.6]

9. Secondary Outcome: Relative Abundance of LY2603618 and the Metabolites of LY2603618 in Feces
Description: as for outcome 8
Time Frame: Day 1 through 7 days postdose
Population: All enrolled participants.
Measure: Mean (Full Range); unit: percentage of [^14C]LY2603618
Arm/Group | [^14C]LY2603618
Number analyzed (Participants) | 3
percentage of [^14C]LY2603618
  LY2603618 (parent) | 5.6 [5.5 to 5.7]
  Metabolites | 61.4 [60.6 to 62.9]

10. Secondary Outcome: The Number of Participants With a Tumor Response
Description: Tumor responses were followed and measured according to Response Evaluation Criteria In Solid Tumors (RECIST) criteria. Complete response was defined as the disappearance of all target and non-target lesions and any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 millimeter (mm) and normalization of tumor marker level of non-target lesions. Partial response was defined as at least a 30% decrease in sum of longest diameter of target lesions. Progressive disease was defined as at least 20% increase in sum of longest diameter of target lesions and minimum 5 mm increase over nadir; Stable disease was defined as small changes that did not meet above criteria.
Time Frame: Baseline through study completion [Cycle 5 (28 days/cycle) and 21-day safety follow-up]
Population: All enrolled participants who had radiological tumor assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Entire Study Population
Number analyzed (Participants) | 2
Participants
  Complete response | 0
  Partial response | 0
  Progressive disease | 2
  Stable disease | 0

ADVERSE EVENTS:
Groups:
- [^14C]LY2603618: Adverse events reported during the first phase of the study. Participants received a single 250 milligram (mg) intravenous dose of LY2603618 containing [^14C]LY2603618 and then completed a minimum 7-day washout period.
- LY2603618 + Gemcitabine: Adverse events reported during the second phase of the study. After completing the first phase [a single 250 milligram (mg) intravenous dose of LY2603618 containing [^14C]LY2603618 followed by a minimum 7-day washout period], participants received Gemcitabine 1000 milligrams per square meter (mg/m^2) administered intravenously on Days 1, 8, and 15 with 230 mg LY2603618 administered intravenously on Days 2, 9 and 16 of a 28-day cycle until unacceptable toxicity or disease progression.
Arm/Group | [^14C]LY2603618 | LY2603618 + Gemcitabine
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | [^14C]LY2603618 (N=3) | LY2603618 + Gemcitabine (N=3)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (3)
Vomiting (Gastrointestinal disorders) | 1 (1) | 3 (5)
Chest discomfort (General disorders) | 0 (0) | 1 (1)
Chills (General disorders) | 1 (1) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0)
Injection site reaction (General disorders) | 1 (1) | 1 (1)
Malaise (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 1 (2)
Pain (General disorders) | 1 (1) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Study stopped early due to low enrollment, therefore data for evaluation was limited. Study not designed for efficacy assessments, however, tumor response data was collected and reported during Continued Access Phase.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days